CLINICAL TRIAL: NCT07293065
Title: A Multicenter, Double-Blinded, Placebo-Controlled Phase III Clinical Trial to Evaluate the Long-term Efficacy of Recombinant Zoster Vaccine (CHO Cell) in Adults Aged 40 Years and Above
Brief Title: Long-term Efficacy of Recombinant Zoster Vaccine (CHO Cell) Study
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: MAXVAX Biotechnology Limited Liability Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: MKKCT-100-005
Record Dates: First submitted 2025-11-20; First posted 2025-12-18 (Actual); Last update posted 2025-12-18 (Actual); Status verified 2025-12

CONDITIONS: Herpes Zoster
MeSH Terms: conditions — Herpes Zoster

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Vaccine Group (Experimental): Subjects will receive Recombinant Zoster Vaccine (CHO cell) according to a 0, 2-month schedule
  Interventions: Biological: Recombinant Zoster Vaccine (CHO Cell)
- Placebo Group (Placebo Comparator): Subjects will receive NaCl solution placebo according to a 0, 2-month schedule
  Interventions: Biological: NaCl solution Placebo

INTERVENTIONS:
Biological: Recombinant Zoster Vaccine (CHO Cell) — 0.5 mL per dose, containing a total of 50 µg recombinant varicella zoster virus glycoprotein E, adjuvanted with MA105. Intramuscular injection
  Arms: Vaccine Group
Biological: NaCl solution Placebo — 0.5 mL per dose, containing 4.5 mg sodium chloride. Intramuscular injection
  Arms: Placebo Group

SUMMARY:
The purpose of the sutdy is to evaluate the protective efficacy of Recombinant Herpes Zoster Vaccine (CHO Cell) (hereinafter referred to as "the investigational vaccine") in preventing herpes zoster at 13-36 months after complete immunization with the 0- and 2-month immunization schedule in individuals aged 40 years and older.

ELIGIBILITY:
Inclusion Criteria:

1. Participants in the MKKCT-100-003 study who have completed two doses of the investigational vaccine;
2. Males or females able to provide legal identity certificate;
3. Participants voluntarily agree to participate in the study, and sign the informed consent form;
4. Able to understand the study procedures and participate in all scheduled follow-up visits, and able to comply with the protocol requirements (such as cooperating in filling out questionnaires/scales, and being regularly contacted during the study for evaluation, etc.).

Exclusion Criteria:

1. Participants who plan to use any products (drugs, vaccines, or medical devices) other than the investigational product for the prevention of VZV infection before signing the informed consent form or during the study period;
2. Participants with a history of herpes zoster;
3. Participants with any confirmed or suspected immunosuppressive or immunodeficiency condition caused by diseases (e.g., malignant tumors, human immunodeficiency virus infections, etc.) or immunosuppressive/cytotoxic treatments (e.g., medications used during cancer chemotherapy, organ transplantation, or treatment of autoimmune diseases);
4. Participants who are currently participating in or plan to participate in other clinical trials during the study;
5. Significant underlying diseases or any other condition that, in the opinion of the investigator, may prevent completion of the trial.

Min Age: 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 12000 (Estimated)
Dates: Start 2025-12-19 (Estimated); Primary Completion 2027-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
The person-year incidence of confirmed herpes zoster cases among individuals aged 40 years and older, 13 to 36 months after completing the full vaccination course with the investigational vaccine according to the 0- and 2-month immunization schedule. | At 13~36 months after the last vaccination
  A suspected case of HZ was confirmed either: by Polymerase Chain Reaction (PCR) or by the Endpoint Adjudication Committee (EAC), consisting of physicians with HZ expertise.

SECONDARY OUTCOMES:
The person-year incidence of confirmed herpes zoster cases among individuals aged 40 years and older: from 30 days to 36 months after completing the full vaccination course, and the annual person-year incidence from 30 days after the full vaccination. | At 30 days~36 months after the last vaccination.
The person-year incidence rate of confirmed Herpes Zoster (HZ) cases during the periods of 30 days to 36 months, 13 to 36 months, and annually after 30 days post full-course immunization, in populations of different age groups. | 30 days to 36 months, 13 to 36 months, and 30 days after the last vaccination.
Incidence of any and severe Postherpetic Neuralgia (PHN) cases per person years in subjects aged 40 years and older, 40-49years , 50-59 years , 60-69 years and ≥70 years , with confirmed HZ. | 30 days after the last vaccination.

CONTACTS AND LOCATIONS:
Locations (4):
- China (4):
  - Hebei Provincial Center for Disease Control and Prevention, Shijiazhuang, Hebei
  - Henan Center for Diseases Control and Prevention, Zhengzhou, Henan
  - Hubei Provincial Center for Disease Control and Prevention, Wuhan, Hubei
  - Yunnan Center For Disease Control and Prevention, Kunming, Yunnan

IPD SHARING:
Plan to Share IPD: No